CLINICAL TRIAL: NCT06817525
Title: Nab-P+Cb+PD1 Inhibitor Neoadjuvant Therapy for Early TNBC: a Single Center, Non Blinded, Randomized Phase II Clinical Trial
Brief Title: Nab-P+Cb+PD1 Inhibitors as Neoadjuvant Therapy for Early TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-020
Record Dates: First submitted 2024-12-05; First posted 2025-02-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Triple-negative Breast Cancer
Keywords: Pathological complete remission rate; Triple-negative breast cancer; Camrelizumab; Neoadjuvant therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6*Chemotherapy drugs(Nab-P, d1, Cb, d1)+6*Immunosuppressants（d1) (Active Comparator): Group A： 6*Albumin-bound paclitaxe (260 mg/m²,d 1)+6*Carboplatin (AUC=5, d 1)+6*Camrelizumab (200 mg, d 1);
  Interventions: Drug: 6*Nab-P (d 1)+6*Cb ( d 1)+6*PD1 (d 1)
- 6*Chemotherapy drugs（Nab-P, d1,8,15, Cb, d1)+6*immunosuppressants（d1, ) (Active Comparator): Group B: 6*Albumin-bound paclitaxe (125 mg/m²,d 1,8,15)+6*Carboplatin (AUC=5, d 1 )+6*Camrelizumab (200 mg, d 1);
  Interventions: Drug: 6*Nab-P (d 1,8,15)+6*Cb ( d 1)+6*PD1 (d 1)

INTERVENTIONS:
Drug: 6*Nab-P (d 1)+6*Cb ( d 1)+6*PD1 (d 1) — This study is a single center, non blinded, randomized phase II clinical trial. A total of 64 TNBC patients are planned to be enrolled. Patients who meet the inclusion criteria will be randomly divided into two groups at a ratio of 1:1 and stratified according to T stage and N stage.
  Group A： Albumin-bound paclitaxe (260 mg/m²,d 1)+Carboplatin (AUC=5, d 1)+Camrelizumab (200 mg, d 1), 21 days as one cycle, 6 cycles;
  Other Names: 6*Albumin-bound paclitaxe (d 1)+6*Carboplatin ( d 1)+6*Camrelizumab (d 1)
  Arms: 6*Chemotherapy drugs(Nab-P, d1, Cb, d1)+6*Immunosuppressants（d1)
Drug: 6*Nab-P (d 1,8,15)+6*Cb ( d 1)+6*PD1 (d 1) — This study is a single center, non blinded, randomized phase II clinical trial. A total of 64 TNBC patients are planned to be enrolled. Patients who meet the inclusion criteria will be randomly divided into two groups at a ratio of 1:1 and stratified according to T stage and N stage.
  Group B: Albumin-bound paclitaxe (125 mg/m²,d 1,8,15)+Carboplatin (AUC=5, d 1 )+Camrelizumab (200 mg, d 1), 21 days as one cycle, 6 cycles;
  Other Names: 6*Albumin-bound paclitaxe (d 1,8,15)+6*Carboplatin ( d 1)+6*Camrelizumab (d 1)
  Arms: 6*Chemotherapy drugs（Nab-P, d1,8,15, Cb, d1)+6*immunosuppressants（d1, )

SUMMARY:
We plan to explore the efficacy and safety of albumin-bound paclitaxel+carboplatin+Camrelizumab in neoadjuvant therapy for early TNBC patients, optimize the administration method and drug combination therapy.

DETAILED DESCRIPTION:
This study is a single center, non blinded, randomized phase II clinical trial. A total of 64 TNBC patients are planned to be enrolled. Patients who meet the inclusion criteria will be randomly divided into two groups (Group A and Group B) at a ratio of 1:1, and stratified according to T stage and N stage. The administration regimen is as follows: Group A： albumin-bound paclitaxe (260 mg/m²,d 1)+Carboplatin (AUC=5, d 1)+Camrelizumab (200 mg, d 1), 21 days as one cycle, 6 cycles; Group B: albumin-bound paclitaxe (125 mg/m²,d 1,8,15)+Carboplatin (AUC=5, d 1 )+Camrelizumab (200 mg, d 1), 21 days as one cycle, 6 cycles

Primary endpoint: Pathological complete response rate (pCR rate).

Secondary study endpoints: Objective response rate (ORR), event free survival rate (EFS), disease-free survival (DFS), distant disease free survival (DDFS), and safety.

Exploratory endpoints: Differences in efficacy and immune microenvironment under different administration methods

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old;
2. Clinically and pathologically confirmed cT2- cT4d, or cT1c with axillary lymph node metastasis;
3. Three negative type and invasive breast cancer confirmed by histopathology;

   Three negative breast cancer is defined as:
   * ER and PR negative (IHC nuclear staining<10%)
   * Her-2 negative (IHC 0, 1+without FISH, or IHC 2+without FISH amplification)
4. Clinically measurable lesions:

   Measurable lesions displayed by ultrasound, mammography, or MR (optional) within one month prior to screening;
5. Organ and bone marrow function tests within 2 weeks before chemotherapy indicate no contraindications for chemotherapy:

   * Absolute value of neutrophil count ≥ 2.0 × 109/L
   * Hemoglobin ≥ 100g/L
   * Platelet count ≥ 100 × 109/L
   * Total bilirubin<1.5 ULN (upper limit of normal)
   * Creatinine<1.5 × ULN
   * AST/ALT < 1.5×ULN；
   * Thyroid stimulating hormone (TSH) ≤ upper limit of normal (ULN); If there are abnormalities, T3 and T4 levels should be examined. If T3 and T4 levels are normal, they can be selected
   * Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN, while meeting international standards Normalization ratio (INR) ≤ 1.5 ULN (not receiving anticoagulant therapy);
6. Cardiac ultrasound EF value ≥ 55%;
7. Women of childbearing age who tested negative for serum pregnancy test 14 days before randomization;
8. ECOG score ≤ 1 point;
9. Voluntary signing of informed consent

Exclusion Criteria:

1. There is evidence of metastatic breast cancer (in order to exclude metastatic breast cancer, chest and abdomen CT and bone scanning should be performed at any time point before diagnosis and randomization; PET/CT scanning can be used as an alternative imaging inspection method);
2. Have Received chemotherapy, endocrine therapy, targeted therapy, radiation therapy, etc. for this disease;
3. The patient has a second primary malignant tumor, in addition to: fully treated skin cancer;
4. Received treatment with anti-PD-1, anti-PDL1, anti-PD-L2 drugs, or other immunotherapy;
5. Diagnosed with immunodeficiency or autoimmune diseases;
6. Severe lung or heart disease;
7. Hepatitis B and C are in active phase;
8. History of organ transplantation or bone marrow transplantation;
9. Pregnant or lactating women;
10. Due to serious and uncontrollable medical conditions, researchers believe there are contraindications to chemotherapy;
11. Screening for clinically significant bleeding symptoms or significant bleeding tendencies within the previous month;
12. Screening for arteriovenous thrombosis events such as deep vein thrombosis and pulmonary embolism that occurred within the previous 3 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response rate(pCR) | through study completion, an average of 1 year
  Pathological Complete Response (pCR) rate: It refers to the absence of any invasive cancer in the resected specimens (breast + axilla) after completion of neoadjuvant chemotherapy and surgery (i.e., ypT0/is, ypN0).

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 24 weeks
  Objective response rate (ORR) based on RECIST v1.1 assessment, defined as the number of target lesion responders evaluated by MRI/ultrasound;
Event-Free Survival (EFS) | 5 years after surgery
  EFS is defined as the time from randomization to any of the following events: disease progression, local or remote recurrence, second primary malignant tumor (breast cancer or other cancers) or death caused by any reason during neoadjuvant treatment;
Disease free survival (DFS) | 5 years after surgery
  DFS is defined as the time from surgery to any of the following events: local or distant recurrence, or death for any reason;
Disease free survival (DDFS) | 5 years after surgery
  The time from surgery to distant recurrence or death for any reason;
Incidence of treatment-emergent adverse events | After each cycle of chemotherapy (21 days as 1 cycle)]
  Evaluate the nature, incidence, and severity of adverse events according to CTCAE 5.0.

OTHER OUTCOMES:
Association of the tumor microenvironment with treatment response | up to 24 weeks
  Multiple immunofluorescence: CD3+CD4+PD1+KI67; CD3+CD8+PD1+KI67; GZMB; TCF-1; CD31; NG-2 in tumor tissue.
Association of peripheral blood lymphocyte subsets and cytokines with treatment response | up to 24 weeks
  Flow cytometric assessment of peripheral blood lymphocyte subsets: CD3+CD4+PD1+KI67; CD3+CD8+PD1+KI67 and Detection of peripheral blood cytokines: vascular endothelial growth factor (VEGF), angiopoietin-2 (ANG-2), basic fibroblast growth factor (bFGF), transforming growth factor-β1 (TGF-β1), and endostatin (ES)

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China